CLINICAL TRIAL: NCT00668876
Title: Effects of Immunonutrition on Surgical Site Infection and Th1/Th2/Th17 Differentiation in Patients Undergoing Pancreaticoduodenectomy
Brief Title: Effects of Immunonutrition in Patients Undergoing Pancreaticoduodenectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chiba University (Other)
Responsible Party: Chiba University, Chiba University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: furukawa2008
Record Dates: First submitted 2008-04-28; First posted 2008-04-29 (Estimated); Last update posted 2008-12-03 (Estimated); Status verified 2008-10

CONDITIONS: Pancreaticoduodenectomy
Keywords: immunonutrition; pancreaticoduodenectomy; Th1; Th2; Th17
MeSH Terms: interventions — Long-Term Synaptic Depression; Parenteral Nutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): Group A: perioperative immunonutrition
  Interventions: Dietary Supplement: Oral IMPACT
- 2 (Active Comparator): Group B: postoperative immunonutrition
  Interventions: Dietary Supplement: Oral IMPACT
- 3 (Active Comparator): Group C: control
  Interventions: Dietary Supplement: Parenteral nutrition

INTERVENTIONS:
Dietary Supplement: Oral IMPACT — oral supplementation for 5 days(1 L/d )before surgery of a formula enriched with arginine, omega-3 fatty acids, and RNA
  Other Names: oral IMPACT; Ajinomoto Pharma Co., Ltd, Tokyo, Japan
  Arms: 1
Dietary Supplement: Oral IMPACT — postoperative enteral infusion of the formula with arginine, omega-3 fatty acids, and RNA
  Arms: 2
Dietary Supplement: Parenteral nutrition — Parenteral nutrition
  Arms: 3

SUMMARY:
The purpose of this study is to determine whether immunonutrition is effective on surgical site infection and Th1/Th2/Th17 differentiation in patients undergoing pancreaticoduodenectomy

DETAILED DESCRIPTION:
Perioperative immunonutrition is reported to improve the incidence of postoperative infectious complication in patients with gastrointestinal surgery. It has also been recognized that Th1/Th2 balance shifts toward Th2 by surgical stress. On the other hand, the change of Th17 status after surgery has not been established. Furthermore, The change of Th1/Th2 balance and Th17 status with immunonutrition on pancreaticoduodenectomy have not been reported yet.

Objective of this study is to investigate the effects of perioperative immunonutrition on incidence of postoperative infectious complication, Th1/Th2 balance and Th17 status after pancreaticoduodenectomy.

ELIGIBILITY:
Inclusion Criteria:

* patients underwent pancreaticoduodenectomy

Exclusion Criteria:

* age younger than 18 years or older than 75 years
* preoperative chemotherapy or radiation
* ongoing infection
* diabetes mellitus
* gastrointestinal obstruction
* respiratory dysfunction
* cardiac dysfunction
* hepatic dysfunction
* renal failure
* history of recent immunosuppressive or immunological diseases
* preoperative evidence of widespread metastatic disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2006-05; Primary Completion 2008-01 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
surgical site infection after surgery | 30days

SECONDARY OUTCOMES:
plasma IL-6, CRP, Th1/Th2 balance, Th17 status | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Daisuke Suzuki, Principal Investigator — Chiba University
Locations (1):
- Chiba University, Chiba, Chiba, Japan